CLINICAL TRIAL: NCT06760403
Title: Investigation of the Efficacy of Hypochlorous Acid as a Postoperative Wound Antiseptic: A Randomized Controlled Pilot Study
Brief Title: Efficacy of Hypochlorous Acid as a Postoperative Wound Antiseptic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Sema Nur Sevinc, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MCT4
Record Dates: First submitted 2024-12-24; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Wound Healing
Keywords: gingival overgrowth; gingivoplasty; gingivectomy; hypochlorous acid; chlorhexidine
MeSH Terms: conditions — Gingival Overgrowth | interventions — Hypochlorous Acid

STUDY DESIGN:
Intervention Model Description: The study included 24 systemically healthy individuals who were randomly divided into three groups: 1) Hypochlorous acid, 2) Chlorhexidine, and 3) Saline.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Hypochlorous Group (Experimental): In the hypochlorous acid group, 15 ml was used as a postoperative gargle, 2 times * 7 days.
  Interventions: Drug: Hypochlorous acid
- Chlorhexidine Group (Active Comparator): In the clorhexidine group, 15 ml was used as a postoperative gargle, 2 times * 7 days.
  Interventions: Drug: Hypochlorous acid
- Saline Group (Placebo Comparator): In the saline group, 15 ml was used as a postoperative gargle, 2 times * 7 days.
  Interventions: Drug: Hypochlorous acid

INTERVENTIONS:
Drug: Hypochlorous acid — Hypochlorous acid, chlorhexidine and saline groups were compared as postoperative gargles after gingivectomy surgery.

SUMMARY:
The aim was to examine the effectiveness of hypochlorous acid on postoperative wound healing in 24 systemically healthy gingivectomy participants aged 12-30. The participants were divided into 3 groups as hypochlorous acid group, chlorhexidine group and saline group and their wound healing was evaluated on the 1st, 3rd and 7th days.

DETAILED DESCRIPTION:
The aim of this study was to investigate the effectiveness of hypochlorous acid on postoperative wound healing in 24 participants aged 12-30 who underwent gingivectomy involving the 6 anterior teeth of the upper or lower jaw with chronic inflammatory gingival overgrowth. The participants were divided into 3 groups as hypochlorous acid group, chlorhexidine group and saline group and were called for control on the 1st, 3rd and 7th days to evaluate wound healing. Periodontal indexes, visual analog scale (VAS), H2O2, plaque staining agent test, and histological analyzes were used to evaluate wound healing. The data were analyzed statistically.

ELIGIBILITY:
Inclusion Criteria:

* Gingival overgrowth affecting at least six teeth symmetrically in the mandibular or maxillary anterior area
* No attachment and bone loss
* 7 days before the surgery, full-mouth plaque index (PI) < 25% and a full-mouth gingival bleeding index (GBI) < 25%.
* the keratinized tissues surrounding the teeth are at least 2 mm wide.

Exclusion Criteria:

* Smoking or alcohol use
* Patients who have undergone systemic antimicrobial therapy and surgical procedures within the last 3 months
* Pregnancy or lactation
* Immunodeficiency or immunosuppressive drug therapy

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Plaque index | Baseline, Day 7
  The amount of plaque was scored.
Gingival index | Baseline, Day 7
  The gingival status was scored.
Probing depth | Baseline, Day 7
  The periodontal pocket depth was performed (mm).
Clinical attachment level | Baseline, Day 7
  The clinical attachment level was measured (mm).
Bleeding on probing | Baseline, Day 7
  The gingival status was scored.(%)
Epithelialization with plaque staining agent | Day 1, 3, and 7
  The wound surface epithelialization was observed with plaque staining agent. The wound surface was stained with plaque staining dye and the dark colored area is calculated as mm2.
Epithelialization with H2O2 | Day 3 and 7
  The wound surface epithelialization was observed with H2O2. Scored as foaming present/absent after application with H2O2
Histological analysis | Day 1, 3, and 7
  Histological analysis evaluated epithelial keratinization, regeneration, and/or degeneration during the healing process and to obtain epithelial samples repeatedly. The number of keratinocytes was counted.
postoperative pain with Visiual Analogue Scale (VAS) | Day 3 and 7
  VAS scores were taken on the 3rd and 7th days without any intervention to the patient. Scored between 1-10 as 1 was no pain, 10 was pain.

CONTACTS AND LOCATIONS:
Overall Officials: Sema Nur Sevinç Gül, Dr., Principal Investigator — Ataturk University
Locations (1):
- Atatürk University Faculty of Dentistry, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burian EA, Sabah L, Kirketerp-Moller K, Gundersen G, Agren MS. Effect of Stabilized Hypochlorous Acid on Re-epithelialization and Bacterial Bioburden in Acute Wounds: A Randomized Controlled Trial in Healthy Volunteers. Acta Derm Venereol. 2022 May 31;102:adv00727. doi: 10.2340/actadv.v102.1624. PMID 35578822